CLINICAL TRIAL: NCT05692674
Title: A Prospective Phase II Study for Adjuvant Hypofractionated Intensity-modulated Proton Radiotherapy for Post Operative Breast Cancer With Implantation Reconstruction
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Proton and Heavy Ion Center (Other)
Responsible Party: Principal Investigator, Qing Zhang,MD, Professor, Shanghai Proton and Heavy Ion Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPHIC-TR-BCa2022-02
Record Dates: First submitted 2023-01-11; First posted 2023-01-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Breast Cancer
Keywords: breast cancer; hypofractionated; proton radiotherapy; implantation reconstruction; postoperative adjuvant radiotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- adjuvant hypofractionated intensity-modulated proton radiotherapy (Experimental): CTV1: chest wall ± regional lymph drainage area, proton therapy.
  Interventions: Radiation: adjuvant hypofractionated intensity-modulated proton radiotherapy

INTERVENTIONS:
Radiation: adjuvant hypofractionated intensity-modulated proton radiotherapy — CTV1: chest wall ± regional lymph drainage area, 40.05Gy (RBE) in 15 fractions with proton radiotherapy;

SUMMARY:
The incidence of breast reconstruction failure after conventional photon radiotherapy for breast cancer is about 18.7%. At present, there is limited data on proton radiotherapy for post operative breast cancer with implantation reconstruction. Proton radiotherapy for breast cancer can significantly reduce the radiation dose of the ipsilateral heart and lung, thereby reducing the incidence of cardiac events and radiation pneumonia. This study is aimed at the study of adjuvant hypofractionated intensity-modulated proton radiotherapy for post operative breast cancer with implantation reconstruction. It can provide an ideal treatment option for such patients to effectively protect the heart and lungs without increasing the failure rate of breast reconstruction after adjuvant radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* 1: Patients with pathologically confirmed breast cancer

  2: Indications: patients who need adjuvant radiotherapy after mastectomy and implant reconstruction

  3: No distant metastasis

  4: Had no chest and breast radiotherapy history

  5: Between the ages of 18 and 80

  6: ECOG general status score is 0-2,There are no serious pulmonary hypertension, cardiovascular disease, peripheral vascular disease, serious chronic heart disease and other complications that may affect the radiotherapy

  7: Non pregnancy (confirmed by serum or urine β- HCG test) or lactating women

  8: The patient must sign the informed consent form for receiving radiotherapy.

Exclusion Criteria:

* 1: No pathological confirmation；

  2: Distant metastasis；

  3: Had chest and breast radiotherapy history

  4: Organs at risk could not achieve safe dose

  5: Pregnancy (confirmed by serum or urine β- HCG test) or lactating women

  6: Poor general health status, i.e. KPS<70, or ECOG>2

  7: There are serious complications that may affect the radiotherapy, including: a) unstable angina, congestive heart failure and myocardial infarction requiring hospitalization in the past 6 months； b) Acute bacterial or systemic fungal infection；c) Chronic obstructive pulmonary disease exacerbation or other respiratory diseases need hospitalization； d) Patients with immunosuppression；e) With connective tissue disease, such as active scleroderma or lupus and other contraindications to radiotherapy；

  8: Unable to understand the purpose of treatment or unwilling/unable to sign informed consent.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2023-01-10 (Estimated); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
the failure rate of breast reconstruction after hypofractionated proton radiotherapy | within 2 years after hypofractionated proton radiotherapy
  Reoperation

SECONDARY OUTCOMES:
Acute and late toxicities | within 5 years after radiotherapy
  Treatment related toxicity assessed by CTCAE v4.03
Tumor local control rate, overall survival rate and progression free survival rate | within 5 years after radiotherapy
  The Ipsilateral breast and regional lymph nodes recurrence, death and progression

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Proton and Heavy Ion center, Shanghai, Shanghai Municipality, China